CLINICAL TRIAL: NCT01957085
Title: Incidence of Undiagnosed Hepatitis C Infection in an Urban Hospital
Brief Title: Undiagnosed Hepatitis C Infection in an Urban Hospital
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Undiagnosed Hepatitis C
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — All leftover sera and plasma will be banked at -70 degrees Celsius in a secure laboratory for potential future research activities
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized Patients: Observation only. All patients admitted to Temple University Hospital on the study day. Observational only, no intervention.
  Interventions: Other: observation only

INTERVENTIONS:
Other: observation only — This is an observational only, nonintervention study. There will be no patient contact. This was a de-identified point prevalence study of hepatitis C infection in hospitalized patients in an inner city hospital.

SUMMARY:
The Centers for Disease Control and Prevention estimates that there are approximately 3.2 million people in the United States infected with hepatitis C and a significant percentage of these patients are unaware of their diagnosis. This study will attempt to determine the point prevalence of undiagnosed hepatitis C infection in an urban hospital population. All patients admitted to the hospital on two separate days will have hepatitis C testing done on leftover serum and plasma that was collected as part of routine inpatient lab work. Our primary goal is to determine the number of undiagnosed hepatitis C infected patients in our hospitalized population. We will also compare these rates to specific demographic characteristics, such as age, race, gender, zip code and type of insurance to see if any associations exist between these demographics and undiagnosed hepatitis C infection.

DETAILED DESCRIPTION:
De-identified study of Hepatitis C infection point prevalence in the inpatient setting of an inner city hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to Temple University Hospital on either of the study dates

Exclusion Criteria:

* Patients admitted on both study dates will only be counted once

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Temple University Hospital on the study dates
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bettiker, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This is a de-identified, observational only study with no intervention. Individual participant data will not be released.

REFERENCES:
- [Background] Ly KN, Xing J, Klevens RM, Jiles RB, Ward JW, Holmberg SD. The increasing burden of mortality from viral hepatitis in the United States between 1999 and 2007. Ann Intern Med. 2012 Feb 21;156(4):271-8. doi: 10.7326/0003-4819-156-4-201202210-00004. PMID 22351712
- [Background] Brady KA, Weiner M, Turner BJ. Undiagnosed hepatitis C on the general medicine and trauma services of two urban hospitals. J Infect. 2009 Jul;59(1):62-9. doi: 10.1016/j.jinf.2009.04.008. Epub 2009 May 3. PMID 19473706
- [Background] Seamon MJ, Ginwalla R, Kulp H, Patel J, Pathak AS, Santora TA, Gaughan JP, Goldberg AJ, Tedaldi EM. HIV and hepatitis in an urban penetrating trauma population: unrecognized and untreated. J Trauma. 2011 Aug;71(2):306-10; discussion 311. doi: 10.1097/TA.0b013e31822178bd. PMID 21825931

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospitalized Patients: All patients admitted to Temple University Hospital on the study day
  Observation only, no intervention: Hepatitis C antibody and RNA measured from leftover sera and plasma from the clinical laboratory
Period: Overall Study
Arm/Group | Hospitalized Patients
Started | 366 (Per Institutional Review Board requirements, exact dates are not to be reported)
Completed | 366 (Per Institutional Review Board, exact dates are not to be reported)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hospitalized Patients: All patients admitted to Temple University Hospital on the study day
  Observation only, no intervention: HCV ab and RNA measured from leftover sera and plasma from the clinical laboratory
Arm/Group | Hospitalized Patients
Number analyzed (Participants) | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 238
  >=65 years | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188
  Male | 178
Race/Ethnicity, Customized [Number; unit: participants] — Participants may have selected more than one category for race/ethnicity, and thus the total in the race category is more than the total participants.
  participants
    African American | 184
    Caucasian | 67
    Latino/a | 84
    Asian | 2
    Other | 14
    Unknown | 19
Region of Enrollment [Number; unit: participants] — Country of residence was not determined. Zip code of residence was taken from hospital records
  participants
    United States | 366
h/o: HIV, Hepatitis C infection, Intravenous drug use, HCV treatment [Number; unit: participants] — This category only counts participants with a particular characteristic. Thus, the total number will be less than the total participants.
  participants
    h/o Human Immunodeficiency Virus Infection | 11
    h/o Hepatitis C Infection | 31
    h/o intravenous drug use | 94
    h/o Hepatitis C treatment | 0

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence of Hepatitis C Infection
Description: The point prevalence of hepatitis C infection in our hospitalized patients will be measured on a single day. All leftover plasma/serum samples will be de-identified and tested for hepatitis C antibody and if antibody positive will be tested for hepatitis C polymerase chain reaction. Results reported as percentage of subjects who are viremic.
Time Frame: Single 24 hour period
Measure: Number; unit: percentage of total subjects
Arm/Group | Hospitalized Patients
Number analyzed (Participants) | 366
percentage of total subjects | 9

2. Other Pre Specified Outcome: Number of Evaluable Participants Age 50 or Older and Point Prevalence of Hepatitis C Viremia
Description: Association between point prevalence of hepatitis C viremia and evaluable participants age 50 or older.
Time Frame: Single 24 hour period
Population: Number of patients with evaluable plasma
Measure: Number; unit: participants
Groups:
- Hospitalized Patients/Participants: All patients admitted to Temple University Hospital on the study day
  Observation only, no intervention: HCV ab and RNA measured from leftover sera and plasma from the clinical laboratory
Arm/Group | Hospitalized Patients/Participants
Number analyzed (Participants) | 237
participants
  # viremic >=50 yrs w h/o HCV | 15
  # viremic >=50 yrs w/o h/o HCV | 9
  Without viremia >=50 yrs | 213
Statistical Analysis 1: Comparison: Hospitalized Patients/Participants; Test type: Superiority or Other; p = .04, Chi-squared — Statistical significance was set at .05 to determine statistical significance

3. Other Pre Specified Outcome: Number of Evaluable Patients With Hepatitis C Viremia by Gender
Description: Association between the incidence of hepatitis C infection and gender.
Time Frame: Single 24 hour period
Population: Number of evaluable patients
Measure: Number; unit: participants
Arm/Group | Hospitalized Patients/Participants
Number analyzed (Participants) | 341
participants
  Viremic females with history of Hepatitis C | 8
  Viremic females without a history of Hepatitis C | 6
  Females without viremia | 165
  Viremic males with history of Hepatitis C | 8
  Viremic males without history of Hepatitis C | 8
  Males without viremia | 146
Statistical Analysis 1: Comparison: Hospitalized Patients/Participants; Test type: Superiority or Other; p > .05, Chi-squared

4. Other Pre Specified Outcome: Number of Patients With Hepatitis C Viremia by Race and Ethnicity
Description: Association between the incidence of hepatitis C infection by race and ethnicity
Time Frame: Single 24 hour period
Population: Number of evaluable patients
Measure: Number; unit: Participants
Arm/Group | Hospitalized Patients/Participants
Number analyzed (Participants) | 341
Participants
  Viremic AA | 14
  Viremic White | 8
  Viremic Latino/a | 8
  Viremic Other/unknown | 1
  Non-viremic AA | 156
  Non-viremic white | 55
  Non-viremic Latino/a | 70
  Non-viremic other/unknown | 29
Statistical Analysis 1: Comparison: Hospitalized Patients/Participants; Test type: Superiority or Other; p > .05, Chi-squared

5. Other Pre Specified Outcome: Association Between Evaluable Viremic Patients and Length of Stay in the Hospital
Description: Association between hepatitis C infection and the patient's length of stay in the hospital.
Time Frame: Single 24 hour period
Population: Length of stay in days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Hospitalized Patients
Number analyzed (Participants) | 341
Days
  Length of stay, viremic patients w h/o HCV | 8 [4 to 12]
  Length of stay, viremic patients w/o h/o HCV | 5.5 [0 to 11.5]
  Length of stay, aviremic patients | 7 [6 to 7]

6. Other Pre Specified Outcome: Number of Evaluable Patients by Prior Visits to the Health System
Description: Number of evaluable patients with at least one prior health system visit in the past 3 years by hepatitis C viremia
Time Frame: Single 24 hour period
Population: Number of evaluable patients
Measure: Number; unit: participants
Arm/Group | Hospitalized Patients
Number analyzed (Participants) | 341
participants
  Viremic patient, h/o HCV with >= 1 prior visit | 14
  Viremic patient, no h/o HCV with >=1 prior visit | 12
  Non-Viremic patient, with >=1 prior visit | 221
  Viremic patient, h/o HCV, no prior visit | 2
  Viremic patient, no h/o HCV, no prior visit | 2
  Non-viremic patient, no prior visit | 90
Statistical Analysis 1: Comparison: Hospitalized Patients; Test type: Superiority or Other; p > .05, Chi-squared

ADVERSE EVENTS:
Time Frame: This was an observation only, no intervention study. There were no adverse advents due to the study.
Arm/Group | Hospitalized Patients
Serious Adverse Events (participants affected / at risk) | 0/366
Other Adverse Events (participants affected / at risk) | 0/366

LIMITATIONS AND CAVEATS:
These results may apply only to inner city, academic medical center hospitals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No